CLINICAL TRIAL: NCT07109973
Title: "Efficacy of a Culturally Adapted Cognitive Behavioral Therapy (CA-CBT) for Depression Among Arab and Asian Adolescents in the United Arab Emirates: A Randomized Controlled Trial"
Brief Title: "Culturally Adapted CBT for Depression in Arab and Asian Adolescents in the UAE (CA-CBT)"
Acronym: CA-CBT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bath Spa University Academic Centre RAK (Other)
Responsible Party: Principal Investigator, Jamal D. Magantor, Program Leader , Department of Psychology, Bath Spa University Academic Centre - RAK, Bath Spa University Academic Centre RAK
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BSU-RAK-PSYCH -2025-0011; BSU-RAK-PSYCH-2025-0011 (Registry Identifier: Ethics Committee Reference Number)
Record Dates: First submitted 2025-07-31; First posted 2025-08-07 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-07

CONDITIONS: Depression; Adolescent Depression; Mental Health; Psychological Stress; Anxiety Disorder
Keywords: Cognitive Behavioural Therapy; Culturally Adapted CBT; Depression; anxiety; Stress
MeSH Terms: conditions — Depression; Psychological Well-Being; Stress, Psychological; Anxiety Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CA-CBT Intervention Group (Experimental): Participants in this group received an 8-week manualized Culturally Adapted Cognitive Behavioural Therapy (CA-CBT) program. Sessions were conducted weekly for 60 minutes by trained therapists with culturally appropriate modifications based on the Southampton Adaptation Framework and the PEN-3 model. Adaptations included religious/spiritual integration, family involvement, and culturally relevant examples.
  Interventions: Behavioral: Culturally Adapted Cognitive Behavioural Therapy (CA-CBT)
- Treatment-as-Usual (TAU) Group (Active Comparator): Participants in this group received standard care as available in their communities. This included access to school counselors, general practitioners, or local mental health clinics. Participants were free to seek or continue any support services of their choice. No structured psychotherapy was administered by the research team.
  Interventions: Other: Treatment-as-Usual (TAU)

INTERVENTIONS:
Behavioral: Culturally Adapted Cognitive Behavioural Therapy (CA-CBT) — CA-CBT is an 8-week manualized therapy program based on core CBT principles, adapted for Arab and Asian adolescents in the UAE. Adaptations followed the Southampton Adaptation Framework (SAF-CaCBT) and the PEN-3 model, including culturally relevant metaphors, integration of religious/spiritual beliefs, family involvement, and emphasis on academic and familial stressors. Sessions were delivered weekly for 60 minutes by trained therapists, with support in English, Arabic, and Tagalog.
  Arms: CA-CBT Intervention Group
Other: Treatment-as-Usual (TAU) — Participants in the TAU group received standard care available within their community. This included optional access to school counselors, general practitioners, or local mental health clinics. No structured psychotherapy or manualized intervention was provided by the research team. This arm served as a pragmatic comparator to evaluate the added value of the Culturally Adapted Cognitive Behavioural Therapy (CA-CBT) intervention.
  Arms: Treatment-as-Usual (TAU) Group

SUMMARY:
This study evaluated the effectiveness of a culturally adapted form of Cognitive Behavioural Therapy (CA-CBT) for reducing depression among Arab and Asian adolescents in the United Arab Emirates (UAE). Depression is a major concern for adolescents in the region, where cultural differences and stigma can make standard mental health treatments less effective.

A total of 175 adolescents aged 13-18, from Filipino, Arab, and other Asian backgrounds, were recruited from schools and communities across the UAE. Participants were randomly assigned to one of two groups: (1) an 8-week CA-CBT program delivered in weekly sessions, or (2) a treatment-as-usual (TAU) group who received available community support.

The CA-CBT program was carefully adapted to reflect the cultural and religious values of participants, including family involvement, use of familiar metaphors, and respect for beliefs about mental illness. The goal was to make therapy more relatable, acceptable, and effective.

The main outcome measured was the severity of depression symptoms before and after the 8-week period. Other outcomes included anxiety, stress levels, and dropout rates. The results showed that CA-CBT significantly reduced depression symptoms more than standard care. The program also had fewer dropouts, meaning more students stayed in therapy.

These findings suggest that adapting evidence-based therapy to reflect cultural values can improve mental health outcomes in diverse communities. The research supports the use of culturally sensitive treatments in school and community mental health programs across multicultural societies like the UAE.

DETAILED DESCRIPTION:
This study was a two-arm, parallel-group, single-blind randomized controlled trial (RCT) conducted to assess the efficacy of a newly developed Culturally Adapted Cognitive Behavioural Therapy (CA-CBT) for adolescent depression in the multicultural context of the UAE. The trial involved 175 adolescents aged 13-18 from Arab, Filipino, and other Asian backgrounds who met the inclusion criteria of scoring ≥10 on the PHQ-A (Patient Health Questionnaire for Adolescents). Participants were randomized to either the CA-CBT intervention group or a treatment-as-usual (TAU) control group.

The CA-CBT group received an 8-week manualized intervention tailored to the cultural values of Arab and Asian adolescents, including content adaptations (e.g., academic and family stress in Filipinos, spiritual concerns in Arabs), process modifications (e.g., family involvement, religious framing), and therapist training. The Southampton Adaptation Framework (SAF-CaCBT) and PEN-3 model guided the cultural adaptation. Sessions were delivered by trained facilitators fluent in English, with support in Arabic and Tagalog.

The TAU group received standard mental health resources as available in the community, including school counselors and primary care services. All participants were assessed at baseline (T0) and after the intervention (T1) using validated tools including PHQ-A for depression and DASS-21 for anxiety and stress.

Primary analysis used a 2 (Group) x 2 (Time) repeated measures ANOVA. Results showed a significant time-by-group interaction, with CA-CBT participants experiencing a greater reduction in depressive symptoms (mean difference = -6.8, p < .001, ηp² = .095) compared to the TAU group. Dropout rates were significantly lower in the CA-CBT group (10.2%) than in the TAU group (19.5%), supporting higher engagement and cultural congruence.

The study protocol received ethical approval from the Bath Spa University Academic Centre RAK IRB (Ref # BSU-RAK-PSYCH-2025-0011) and was registered prospectively (ISRCTN14751844).

The findings demonstrate that CA-CBT is a culturally valid and effective intervention for adolescent depression in diverse populations and support the integration of culturally tailored therapies in school and community-based mental health care systems.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents aged 13 to 18 years old
* Screening positive for mild to moderate depressive symptoms based on the PHQ-9
* Able to understand and communicate in English, Arabic, or Tagalog
* Parental/guardian consent and participant assent provided
* Willing to attend all 8 weekly therapy sessions

Exclusion Criteria:

* Currently undergoing structured psychotherapy or psychiatric treatment
* Diagnosed with severe mental disorders (e.g., psychosis, bipolar disorder)
* Active suicidal ideation requiring emergency intervention
* Significant cognitive or developmental delays that impede participation
* Unwilling or unable to commit to full program attendance

Exclusion Criteria:

-

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 175 (Actual)
Dates: Start 2024-06-15 (Actual); Primary Completion 2025-01-20 (Actual); Study Completion 2025-04-20 (Actual)

PRIMARY OUTCOMES:
Change in depressive symptoms measured by the PHQ-9 scale | Baseline and post-intervention (8 weeks)
  The Patient Health Questionnaire-9 (PHQ-9) will be used to assess the severity of depressive symptoms. Scores range from 0 to 27, with higher scores indicating greater depressive symptom severity. The PHQ-9 is a validated and widely used self-report tool.

CONTACTS AND LOCATIONS:
Locations (1):
- Bath Spa University Academic Centre - Ras Al Khaimah, Ras al-Khaimah, United Arab Emirates, United Arab Emirates

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rathod S, Gega L, Degnan A, et al. The current state of culturally adapted mental health interventions: a meta-review of meta-analyses. Psychol Med. 2018;48(11):1868-1877. doi:10.1017/S0033291717003212
- [Background] Airhihenbuwa CO. Health and Culture: Beyond the Western Paradigm. Thousand Oaks: Sage Publications; 1995.
- [Background] Hinton DE, Jalal B, Weiss MG. Cultural adaptation of cognitive behavioral therapy (CBT). Transcult Psychiatry. 2016;53(6):683-706. doi:10.1177/1363461516678326